CLINICAL TRIAL: NCT04463381
Title: Impact of Choledochotomy Techniques During Laparoscopic CBD Exploration on Short- and Long-term Clinical Outcomes: Time to Change Concepts
Brief Title: Choledochotomy Techniques During LCBDE
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Emad Ali Ahmed Ali, Principal investigator, Sohag University
Other Study IDs: 22/05/2020
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Choledocholithiasis
Keywords: choledochotomy technique; CBD stones; choledocholithiasis
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Group 1: sharp choledochotomy by a scalpel or scissor
  Interventions: Procedure: choledochotomy techniques during LCBDE
- Group 2: choledochotomy by a diathermy hook
  Interventions: Procedure: choledochotomy techniques during LCBDE
- Group 3: choledochotomy by an ultrasonic device
  Interventions: Procedure: choledochotomy techniques during LCBDE

INTERVENTIONS:
Procedure: choledochotomy techniques during LCBDE

SUMMARY:
complications after laparoscopic common bile duct exploration (LCBDE) regarding the choledochotomy technique have not been adequately studied in the literature. Therefore, this study aimed to retrospectively analyze and compare the impact of choledochotomy techniques during LCBDE among patients with choledocholithiasis during the early and late postoperative periods.

DETAILED DESCRIPTION:
Background: complications after laparoscopic common bile duct exploration (LCBDE) regarding the choledochotomy technique have not been adequately studied in the literature. Therefore, this study aimed to retrospectively analyze and compare the impact of choledochotomy techniques during LCBDE among patients with choledocholithiasis during the early and late postoperative periods.

Methods: from March 2014 to February 2018, 85 patients with choledocholithiasis (52 females and 33 males) were enrolled in this study. These patients were treated by LCBDE using various choledochotomy techniques, including scalpel or scissor (28 patients, 33%) in group I, using diathermy hook (35 patients, 41%) in group II, or using an ultrasonic device (22 patients, 26 %) in group III. Postoperative follow-up was done for assessment of all possible complications either early (within 3-6 months postoperatively), or late (2-6 years postoperatively) with meticulous observation and study of any relevant postoperative event.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with choledocholithiasis who underwent LCBDE combined with LC were enrolled in this study. No limitations as regards the stone sizes or numbers were considered. The CBD diameter should be at least ± 1 cm.

Exclusion Criteria:

* Exclusion criteria were normal caliber or stenosed CBD, or the presence of overt cholangitis. Additionally, treated patients with the trans-cystic approach for stone extraction were excluded from this study.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: During the study period, 85 patients (52 females and 33 males) were enrolled in this study which they were complaining of manifestations of CBD stones and treated using laparoscopic approaches, using various choledochotomy techniques.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
biliary leakage/fistula | first postoperative 6 months up to 6 years postoperatively
  According to the international study group of liver surgery, bile leakage is defined as fluid with an elevated bilirubin level (3 times higher than the serum bilirubin measured at the same time) in the abdominal drain or the intra-abdominal fluid on or after POD 3, or as the need for radiologic intervention because of biliary collections or re-laparotomy resulting from biliary peritonitis
biliary stricture | 2-6 years
  The biliary stricture is known as abnormal narrowing of the bile duct associated with the rising of cholestasis indexes. Additionally, it has required an invasive treatment such as ERCP, percutaneous transhepatic drainage, or re-surgery [16]. Biliary complications were diagnosed by trans-tubal cholangiography or through MRCP and could be managed conservatively, ERCP, if there is an accessible route, PTD or surgical intervention.

SECONDARY OUTCOMES:
operative time | from incision to closure
  from incision to closure
intraoperative bleeding | during surgery
  in mm
conversion rate | during surgery
  from laparoscopy to open
jaundice | 2-6 years
  missed stone
wound sepsis | 2-6 years
  infection of the wound
cholangitis | 2-6 years
  inflammation of the biliary system
wound dehiscence | 2-6 years
  Gapped wound
Peritoneal sepsis and abscess | first postoperative 6 months
  peritonitis
Recurrent stones | 2-6 years
  recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Emad Ali Ahmed, MD, PhD, Principal Investigator — Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided